CLINICAL TRIAL: NCT00017030
Title: Phase II Study of ET-743 Given as a Three Hour Intravenous Infusion in Patients With Advanced and/or Metastatic Soft Tissue Sarcoma Previously Treated With Chemotherapy
Brief Title: Ecteinascidin 743 in Treating Patients With Unresectable Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: PMAR-ET-B-022-00; MSKCC-01018; CDR0000068643 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1948
Record Dates: First submitted 2001-06-06; First posted 2004-03-11 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-12

CONDITIONS: Sarcoma
Keywords: stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

INTERVENTIONS:
Drug: trabectedin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ecteinascidin 743 in treating patients who have unresectable advanced or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rate of clinical benefit, in terms of the incidence of objective partial and complete response, stable disease, or minor response of more than 3 months duration, in patients with previously treated, unresectable advanced or metastatic soft tissue sarcoma treated with ecteinascidin 743. II. Determine the progression-free survival, overall survival, and response duration in patients treated with this drug. III. Determine the toxicity profile of this drug in these patients. IV. Determine the pharmacokinetic-pharmacodynamic relationship of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to number of prior cytotoxic therapies for advanced disease (1-2 vs more than 2). Patients receive ecteinascidin 743 IV over 3 hours on day 1. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 36-76 patients (18-38 per stratum) will be accrued for this study within 13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced or metastatic soft tissue sarcoma Unresectable disease Previously treated with at least 1 prior non-adjuvant chemotherapy regimen for advanced or metastatic disease Adjuvant chemotherapy considered first-line treatment for advanced disease if the first relapse is less than 6 months after completion of therapy At least 1 bidimensionally measurable non-irradiated lesion At least 20 mm in at least 1 diameter by CT scan At least 20 by 20 mm for clinically measurable lesion No gastrointestinal stromal sarcoma No HIV-related Kaposi's sarcoma No malignant mesothelioma No chondrosarcomas No symptomatic brain or leptomeningeal involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 OR Karnofsky 60-100% Life expectancy: At least 3 months Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) Alkaline phosphatase no greater than ULN (unless suspected bone metastases present) AST/ALT less than 2.5 times ULN Albumin at least 2.5 g/dL No chronic active liver disease Renal: Creatinine no greater than 1.8 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No congestive heart failure No angina pectoris, even if medically controlled No myocardial infarction within the past year No uncontrolled arterial hypertension or arrhythmias Other: No other neoplastic disease within the past 5 years except non-melanoma skin cancer or carcinoma in situ No other serious illness or medical condition No active infection No history of significant neurological or psychiatric disorders No symptomatic peripheral neuropathy grade 2 or greater Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 1 month after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Recovered from prior immunotherapy No concurrent prophylactic colony-stimulating factors (e.g., filgrastim (G- CSF) or sargramostim (GM-CSF)) during first course of study No concurrent anticancer immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered No other concurrent chemotherapy Endocrine therapy: No concurrent anticancer hormonal therapy Radiotherapy: See Disease Characteristics Recovered from radiotherapy No concurrent radiotherapy except palliative local radiotherapy Surgery: See Disease Characteristics Other: At least 30 days since prior investigational drugs No other concurrent investigational or experimental anticancer drugs No concurrent participation in other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2003-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York